CLINICAL TRIAL: NCT06402565
Title: A Randomized, Controlled, Evaluator-Blinded Study to Assess the Safety and Efficacy of NOX1416 in the Treatment of Chronic, Non-Healing, Diabetic Foot Ulcers
Brief Title: NOX1416 in Treatment of Chronic Non-Healing Diabetic Foot Ulcers
Acronym: NTCDU
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NOxy Health Products, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NO-003
Record Dates: First submitted 2024-04-23; First posted 2024-05-07 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: A total of 40 subjects (25 in the treatment group and 15 in the control group) will be randomized to receive either NOX1416 + SOC or SOC alone.
Who Masked: Outcomes Assessor
Masking Description: Evaluator-Blinded Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NOX1416 and SOC (Experimental): NOX1416 is a foam based gaseous nitric oxide (NO) product that will be topically applied directly onto the wound bed and left on the wound bed for a 5-minute period. Subjects randomized to the NOX1416 treatment group will receive once a day application, for a total of 12 weeks with a double treatment, 10 minutes apart, on the first day.
  Standard of care will include evaluation to document, offloading, adequate arterial flow, wound cleansing, removal of necrotic, infected and/or nonviable tissue by debridement, maintenance of a moist wound environment, and management of infection.
  Interventions: Drug: NOX1416 and SOC
- SOC (Standard of care) (Active Comparator): Subjects randomized to the control group will receive standard of care, alone. Standard of care will include evaluation to document, offloading, adequate arterial flow, wound cleansing, removal of necrotic, infected and/or nonviable tissue by debridement, maintenance of a moist wound environment, and management of infection.
  Interventions: Procedure: SOC (Standard of care)

INTERVENTIONS:
Drug: NOX1416 and SOC — Topical Nitric Oxide
  Other Names: ADVANOX
  Arms: NOX1416 and SOC
Procedure: SOC (Standard of care) — SOC as provided in the Arm/Group description.
  Arms: SOC (Standard of care)

SUMMARY:
The goal of this multi-center, randomized, controlled, evaluator-blinded study is to assess and measure the safety and efficacy of NOX1416 as an adjunct to standard of care (SOC) in the treatment of chronic, non-healing, diabetic foot ulcers (DFUs). Subjects will be randomized to receive treatment with NOX1416 as an adjunct to Standard of Care (SOC) or SOC alone.

The primary objective of the study is to demonstrate the safety and tolerability of NOX1416 as adjunct to SOC. The secondary objective of the study is to evaluate the clinical benefit of daily NOX1416, as an adjunct to SOC, in the treatment of chronic, non-healing diabetic foot ulcers. The study will use a centralized blinded assessor. The blinded assessor will be responsible for assessing the efficacy endpoints such as wound measurements and complete wound closure. The blinded assessor will not be involved in the clinical care of the subject.

DETAILED DESCRIPTION:
A total of 40 subjects (25 in the treatment group and 15 in the control group) will be randomized to receive either NOX1416 plus SOC or SOC alone. NOX1416 is a foam based gaseous nitric oxide (NO) product where NO is delivered topically through a microbubble foam. One pump each of Solution A (0.3g, containing citric acid) and Solution B (0.3g, containing Sodium nitrite) will be dispensed and mixed upon depression of the wye nozzle dispenser, and then applied immediately per each square centimeter of wound area using any sterile applicator. NOX1416 is topically applied directly onto the wound bed and left on the wound bed for a 5-minute period then rinsed off or wiped off with a wet, sterile cloth.

Subjects randomized to the NOX1416 treatment group will receive once a day application, for a total of 12 weeks with a double treatment, 10 minutes apart, on the first day. Subjects randomized to the control group will receive standard of care, alone. Standard of care will include evaluation to document, offloading, adequate arterial flow, wound cleansing, removal of necrotic, infected and/or nonviable tissue by debridement, maintenance of a moist wound environment, and management of infection.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for enrollment in the study only if they meet ALL the following criteria at time of Screening:

1. Male or female subjects aged 18 to 80 years (inclusive) with Type 1 or Type 2 diabetes requiring treatment with oral medications and/or insulin replacement therapy
2. Subject has a glycosylated hemoglobin, HbA1c ≤ 12%. Note: Prior documented HbA1c within the last 3 months of the Screening Visit is acceptable.
3. Presence of at least one diabetic foot ulcer that meets all of the following criteria:

   1. A full-thickness ulcer of University of Texas Wound Classification (UTWCS) Grade IA or IIA
   2. At least 50% of the ulcer is located below the malleoli
   3. Ulcer size (area) is ≥ 1 cm2 and ≤ 10 cm2 (post-debridement at time of randomization)
   4. Unresponsive to standard ulcer care for ≥ 4 weeks (at time of screening)
   5. There is a minimum 1 cm margin between the qualifying Target Ulcer and any other ulcers on the specified foot, post-debridement)
   6. No exposed bone and no tunneling, undermining, or sinus tracts
   7. The index ulcer has a clean base and is free of necrotic debris at time of placement of treatment product.
   8. Index ulcer and/or index ulcer limb may have had prior infection, but infection(s) must be adequately treated and controlled as defined by IDSA Guidelines Grade level 1.
   9. Ulcer must be non-healing as defined as < 25% reduction in size in response to standard of care during the two-week run-in Screening Period (between the first Screening Visit and Baseline) Note: Criterion 3(i) will be evaluated at the time of randomization. If the subject has more than one qualifying diabetic foot ulcer, the ulcer designated as the Target Ulcer will be at the discretion of the Investigator.
4. Adequate circulation to the affected foot as demonstrated by a dorsum transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 30 mmHg or an ABI between 0.7 and ≤ 1.3, or TBI of >0.6 within 3 months of the first Screening Visit. The assessment may also be performed between SV1 and SV2.
5. Subject does not smoke or use tobacco products.
6. Subject, if female of child-bearing potential, has a negative urine pregnancy test at screening, must not be breastfeeding, and willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence) throughout the study.
7. Subject is able and willing to comply with study procedures and applicable dressing changes.
8. Subject demonstrates cognitive and physical ability to administer the treatment as determined by the clinician. If a caregiver will administer the treatment, the caregiver must demonstrate cognitive and physical ability.
9. The index ulcer has been offloaded with protocol defined offloading device throughout the study run-in period for at least 14 days prior to randomization (Run- in period defined as Screening through TV1/Randomization).
10. A signed and dated informed consent form has been obtained from the subject.

Exclusion Criteria:

Subjects meeting ANY of the following criteria at time of Screening will be excluded from enrollment:

1. Ulcers with exposed bone or associated with osteomyelitis. Note: Osteomyelitis should be ruled out by clinical examination (probing of the wound) or X-ray findings, if necessary, by the Investigator.
2. Subject has ulcers secondary to a disease other than diabetes, e.g., fungal ulcerations, malignant ulcerations, and ulcerations due to venous or arterial insufficiency, or due to hematological disorders, in the opinion of the Principal Investigator.
3. Ulcer, which in the opinion of the Investigator, is suspicious for cancer.
4. Subjects with a gangrenous or ischemic toe that may need to be amputated in the opinion of the Investigator.
5. Body mass index (BMI) > 40kg/m2
6. Methemoglobin > 5% at SV1
7. Laboratory values at Screening of:

   * Hemoglobin < 8.5 g/dL
   * White Blood Cells (WBC) < 3.0 X 109 cells/L and > 11 x 109 cells/L
   * Liver function studies [Total bilirubin, aspartate aminotransferase (AST) and alanine transaminase (ALT)] > 3x the upper limit of normal
   * Albumin < 2.5 g/dL
   * Renal function studies [Estimated Glomerular Filtration Rate] < 45
8. Presence of any clinically significant medical condition(s) that, in the opinion of the Investigator, could interfere with wound healing, including but not limited to the following:

   * Vasculitis or connective tissue disease
   * Buerger's disease, Raynaud's or other peripheral vascular disease.
   * Clinically significant claudication or peripheral edema on the affected limb
   * Acute or unstable Charcot foot
   * Aplastic anemia or sickle cell anemia
   * Current sepsis
9. Past or present malignancy below the knee on the same limb as the Target Ulcer;
10. History of radiation at the Target Ulcer site.
11. Subject is currently receiving (i.e., within 30 days of T1 visit) or scheduled to receive any of following medication or therapies during the course of the study.

    * Immunosuppressants (including chronic systemic corticosteroids)
    * Cytotoxic chemotherapy
    * Cytostatic therapy
    * Lower limb revascularization surgery (e.g., angioplasty, artery bypass surgery,)
    * application of bioengineered tissue or skin substitutes
    * use of any investigational drug(s)
12. Subjects who have previously received NOX1416 treatment
13. Subject is unable to comply with offloading device.
14. Revascularization surgery on the lower extremity on which the index ulcer is located within 30 days of Screening Visit (SV1).
15. Has a known hypersensitivity to any of the investigational drug components
16. Subject is susceptible to hemorrhaging or has a congenital or acquired predisposition to hemorrhaging.
17. Subject has a history of self-harm or suicidal ideation.
18. Any reason that the subjects may need to be admitted to inpatient acute care in the opinion of the Investigator.
19. Has any other factor which may, in the opinion of the investigator, compromise participation and/or follow-up in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with a Methemoglobin >5% at any assessment point | 14 weeks
  Methemoglobin is measured using co-oximetry
Incidence and severity of treatment-emergent adverse events (TEAEs) | 16 weeks
  Incidence and severity of treatment-emergent adverse events (TEAEs), including serious adverse events and adverse events resulting in permanent discontinuation of protocol-defined therapy

SECONDARY OUTCOMES:
Proportion of subjects with complete wound closure during the 12 weeks of the Treatment Phase | 12 weeks
  Complete wound closure is defined as 100% re-epithelialization without drainage or dressing requirements confirmed at two consecutive study visits 2 weeks apart. Complete wound closure will be evaluated by the blinded evaluator.
Wound Area Change (%) during the 12 weeks of the Treatment Phase | 12 weeks
  Wound area change is defined as the percentage of wound area change as measured by Swift Imaging device.
Wound volume change (%) during the 12 weeks of the Treatment Phase | 12 weeks
  Wound volume change is defined as the percentage of change based on manual measurements of L x W x D in centimeters.
Time to complete wound closure during the 12 weeks of the Treatment Phase | 12 weeks
  Complete wound closure is defined as 100% re-epithelialization without drainage or dressing requirements confirmed at two consecutive study visits 2 weeks apart. Complete wound closure will be evaluated by the blinded evaluator.
Proportion of subjects who do not develop an infection during the 12 weeks of the Treatment Phase | 12 weeks
  Based on the clinical signs of infection per PI clinical judgement
Changes in Wound-Q Health-Related Quality of Life (Life Impact Psychological, Social) scores during the 12 weeks of the Treatment Phase | 12 weeks
  Life Impact (8 item), Psychological (10 item), and Social (5 item) scales will be used to assess the impact of wound healing on the subject's Quality of Life. There is no overall or total WOUND-Q score. The WOUND-Q is composed of independently functioning scales that are scored separately. To score a scale, the raw scores for the set of items in a scale are added together to produce a total raw score. If missing data is less than 50% of the scale's items, the within person mean for the completed items can be imputed for the missing items prior to computing a total raw score. Once a total raw score for the scale is computed, the Conversion Table can be used to convert the raw score into a score that ranges from 0 (worst) to 100 (best). Higher scores for WOUND-Q scales reflect a better outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Prohealth Research Center, Doral, Florida
  - Family First Medical Research Center, Hialeah Gardens, Florida

IPD SHARING:
Plan to Share IPD: No